CLINICAL TRIAL: NCT04154969
Title: The Effect of Vestibulo-ocular Reflex Improving Exercise on Gait and Balance Among Post Stroke Sub Acute Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Dan Justo (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Dan Justo, Prof. Dan Justo, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-19-6371-DJ-CTIL
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Stroke
Keywords: balance; gait; post stroke rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): daily physiotherapy session as part of the rehab plan, which includes 10 minutes of vestibular exercize.
  Interventions: Other: Physiotherapy including Vestibular rehabilitation
- control (Active Comparator): daily physiotherapy session as part of the rehab plan
  Interventions: Other: conventional Physiotherapy

INTERVENTIONS:
Other: Physiotherapy including Vestibular rehabilitation — vestibular exercise (VOR TX1)
  Arms: intervention
Other: conventional Physiotherapy — conventional Physiotherapy
  Arms: control

SUMMARY:
This study evaluate the effect of Vestibular rehabilitation program as part of physical therapy during rehabilitation post stroke. half of participants will receive vestibular exercise as part of the physiotherpy session, while the other half will receive a conservative physiotherapy session.

DETAILED DESCRIPTION:
Background Stroke global incidence is rising, in Israel 40% of the stroke patients are in need for hospitalized rehabilitation. Improving mobility, and in particular walking after stroke, is utterly important to reduce the risk of falling and is strongly correlated to higher patient autonomy and improved quality of life. During walking balance maintenance, is a complex function relying upon three modalities of sensory information. The sensory weighting process is compromised in stroke patients, so they are excessively reliant on visual information to control their posture. applying vestibular inputs, such as vestibulo-ocular reflex (VOR) habituation exercise, as part of vestibular focused rehabilitation (VR) is one of the methods to trigger sensory reweighting processes in post stroke patients. The VOR role in balance is to assist stabilizing images on the retina during head movement. It may be possible to explain the phenomena of head stabilization during gait in post stroke patients, as an attempt to maintain gaze stability due to reduced dynamic visual acuity (DVA) arising from decreased VOR function.

Aims The aims of this study are firstly to investigate the effectiveness of VOR exercise on gait speed and balance in post stroke patients with no dizziness, and secondly, to test the correlation between the efficiency of the VOR, as reflected by DVA and gait velocity.

Methods A prospective experimental study, randomized controlled, double blinded (assessor and statistician). Sixty adults, 65 years and older, hospitalized in the geriatric rehabilitation departments at the Sheba Medical Center, Israel will be divided to control and intervention groups. The intervention will include physiotherapy sessions including 10 minutes dedicated to VOR habituation exercise, comparing to physiotherapy sessions with no VOR exercise.

Prior to the baseline testing (T1), the participants will perform the outcome measures tests twice (two consecutive days) to determine the smallest real difference. Following this, the outcome measures will be tested at three time-points: before the beginning of the vestibular training (T1); three weeks later, at the termination of the vestibular training (T2) and three weeks after the termination of the training period (T3), to measure retention. For assessing gait and balance, the Dynamic Gait Index (appendix 1), the 10 Meters Walking Test (appendix 2) and the Timed Up and Go test (appendix 3) will be utilized. For assessing balance confidence the Activities-specific Balance Confidence Scale (ABC) questionnaire will be applied. For assessing the DVA, the Dynamic visual acuity test will be applied.

ELIGIBILITY:
Inclusion Criteria:

within 0-3 months of a stroke (ischemic or hemorrhagic; anterior or posterior circulation; not vertebro-basilar stroke).

Exclusion Criteria:

any significant medical illness or blood pressure at rest>110/200 mmHg; a Mini-Mental State Exam score <24, global; a receptive aphasia or an inability to follow 2-point commands; unable to walk 16 meters with no physical assistance.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-10 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Dynamic Gait Index | 10 minute
  scoring walking while performing deferent tasks, such as walking around obstacle, turn head while walking.
10 Meters Walking Test | 1 minute
  timing walking 10 meters walking
Timed Up and Go test | 1 minute
  getting up from a chair, walk for 3 meters and back to the chair.
Activities-specific Balance Confidence Scale | 5 minute
  questionnaire for balance confidence in deferent daily tasks
Dynamic visual acuity test | 5 minute
  assessing the Vestibulo-ocular reflex by quantifying the visual acuity during head movement

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2016 DALYs and HALE Collaborators. Global, regional, and national disability-adjusted life-years (DALYs) for 333 diseases and injuries and healthy life expectancy (HALE) for 195 countries and territories, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1260-1344. doi: 10.1016/S0140-6736(17)32130-X. PMID 28919118
- [Background] ICDC. Stroke Registry Report for 2015-2016.; 2016. https://www.health.gov.il/publicationsfiles/stroke_registry_report_2014-2015.pdf.
- [Background] Ifrah A, Arditi T, Sever L, Tanne D, Koton S. National acute stroke israeli survey (NASIS) 2010. Natl Acute Stroke Isr Surv 2010. 2010;(ICDC):1-43.
- [Background] Tramontano M, Martino Cinnera A, Manzari L, Tozzi FF, Caltagirone C, Morone G, Pompa A, Grasso MG. Vestibular rehabilitation has positive effects on balance, fatigue and activities of daily living in highly disabled multiple sclerosis people: A preliminary randomized controlled trial. Restor Neurol Neurosci. 2018;36(6):709-718. doi: 10.3233/RNN-180850. PMID 30412513
- [Background] Studenski S, Perera S, Patel K, Rosano C, Faulkner K, Inzitari M, Brach J, Chandler J, Cawthon P, Connor EB, Nevitt M, Visser M, Kritchevsky S, Badinelli S, Harris T, Newman AB, Cauley J, Ferrucci L, Guralnik J. Gait speed and survival in older adults. JAMA. 2011 Jan 5;305(1):50-8. doi: 10.1001/jama.2010.1923. PMID 21205966
- [Background] Bonan IV, Marquer A, Eskiizmirliler S, Yelnik AP, Vidal PP. Sensory reweighting in controls and stroke patients. Clin Neurophysiol. 2013 Apr;124(4):713-22. doi: 10.1016/j.clinph.2012.09.019. Epub 2012 Oct 22. PMID 23088814
- [Background] Geurts AC, de Haart M, van Nes IJ, Duysens J. A review of standing balance recovery from stroke. Gait Posture. 2005 Nov;22(3):267-81. doi: 10.1016/j.gaitpost.2004.10.002. Epub 2004 Dec 7. PMID 16214666
- [Background] Sober SJ, Sabes PN. Flexible strategies for sensory integration during motor planning. Nat Neurosci. 2005 Apr;8(4):490-7. doi: 10.1038/nn1427. Epub 2005 Mar 27. PMID 15793578
- [Background] Keshner EA, Kenyon RV, Langston J. Postural responses exhibit multisensory dependencies with discordant visual and support surface motion. J Vestib Res. 2004;14(4):307-19. PMID 15328445
- [Background] Keshner EA, Kenyon RV. The influence of an immersive virtual environment on the segmental organization of postural stabilizing responses. J Vestib Res. 2000;10(4-5):207-19. PMID 11354434
- [Background] Ferre ER, Walther LE, Haggard P. Multisensory interactions between vestibular, visual and somatosensory signals. PLoS One. 2015 Apr 13;10(4):e0124573. doi: 10.1371/journal.pone.0124573. eCollection 2015. PMID 25875819
- [Background] Bonan IV, Colle FM, Guichard JP, Vicaut E, Eisenfisz M, Tran Ba Huy P, Yelnik AP. Reliance on visual information after stroke. Part I: Balance on dynamic posturography. Arch Phys Med Rehabil. 2004 Feb;85(2):268-73. doi: 10.1016/j.apmr.2003.06.017. PMID 14966712
- [Background] Ferre ER, Day BL, Bottini G, Haggard P. How the vestibular system interacts with somatosensory perception: a sham-controlled study with galvanic vestibular stimulation. Neurosci Lett. 2013 Aug 29;550(100):35-40. doi: 10.1016/j.neulet.2013.06.046. Epub 2013 Jul 1. PMID 23827220
- [Background] Tramontano M, Bergamini E, Iosa M, Belluscio V, Vannozzi G, Morone G. Vestibular rehabilitation training in patients with subacute stroke: A preliminary randomized controlled trial. NeuroRehabilitation. 2018;43(2):247-254. doi: 10.3233/NRE-182427. PMID 30040765
- [Background] Clendaniel RA. The effects of habituation and gaze stability exercises in the treatment of unilateral vestibular hypofunction: a preliminary results. J Neurol Phys Ther. 2010 Jun;34(2):111-6. doi: 10.1097/NPT.0b013e3181deca01. PMID 20588098
- [Background] Balci BD, Akdal G, Yaka E, Angin S. Vestibular rehabilitation in acute central vestibulopathy: a randomized controlled trial. J Vestib Res. 2013;23(4-5):259-67. doi: 10.3233/VES-130491. PMID 24284606
- [Background] Yeole UL, Raut RV. Effect of proprioceptive exercise program versus vestibular rehabilitation therapy on risk of fall in elderly. 2018;3(December):117-122.
- [Background] Maas EF, Huebner WP, Seidman SH, Leigh RJ. Behavior of human horizontal vestibulo-ocular reflex in response to high-acceleration stimuli. Brain Res. 1989 Oct 9;499(1):153-6. doi: 10.1016/0006-8993(89)91145-1. PMID 2804663
- [Background] Grossman GE, Leigh RJ, Bruce EN, Huebner WP, Lanska DJ. Performance of the human vestibuloocular reflex during locomotion. J Neurophysiol. 1989 Jul;62(1):264-72. doi: 10.1152/jn.1989.62.1.264. PMID 2754477
- [Background] Lamontagne A, Fung J. Gaze and postural reorientation in the control of locomotor steering after stroke. Neurorehabil Neural Repair. 2009 Mar-Apr;23(3):256-66. doi: 10.1177/1545968308324549. Epub 2008 Dec 5. PMID 19060133
- [Background] Marchetti GF, Whitney SL, Blatt PJ, Morris LO, Vance JM. Temporal and spatial characteristics of gait during performance of the Dynamic Gait Index in people with and people without balance or vestibular disorders. Phys Ther. 2008 May;88(5):640-51. doi: 10.2522/ptj.20070130. Epub 2008 Feb 21. PMID 18292216
- [Background] Mitsutake T, Sakamoto M, Ueta K, Oka S, Horikawa E. Effects of vestibular rehabilitation on gait performance in poststroke patients: a pilot randomized controlled trial. Int J Rehabil Res. 2017 Sep;40(3):240-245. doi: 10.1097/MRR.0000000000000234. PMID 28542112
- [Background] Grossman GE, Leigh RJ, Abel LA, Lanska DJ, Thurston SE. Frequency and velocity of rotational head perturbations during locomotion. Exp Brain Res. 1988;70(3):470-6. doi: 10.1007/BF00247595. PMID 3384048
- [Background] Scheffer AC, Schuurmans MJ, van Dijk N, van der Hooft T, de Rooij SE. Fear of falling: measurement strategy, prevalence, risk factors and consequences among older persons. Age Ageing. 2008 Jan;37(1):19-24. doi: 10.1093/ageing/afm169. PMID 18194967
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Bohannon RW. Comfortable and maximum walking speed of adults aged 20-79 years: reference values and determinants. Age Ageing. 1997 Jan;26(1):15-9. doi: 10.1093/ageing/26.1.15. PMID 9143432
- [Background] Longridge NS, Mallinson AI. The dynamic illegible E-test. A technique for assessing the vestibulo-ocular reflex. Acta Otolaryngol. 1987 Mar-Apr;103(3-4):273-9. PMID 3577760
- [Background] Verbecque E, Van Criekinge T, Vanloot D, Coeckelbergh T, Van de Heyning P, Hallemans A, Vereeck L. Dynamic Visual Acuity test while walking or running on treadmill: Reliability and normative data. Gait Posture. 2018 Sep;65:137-142. doi: 10.1016/j.gaitpost.2018.07.166. Epub 2018 Jul 19. PMID 30558920